CLINICAL TRIAL: NCT01450215
Title: Randomized Trial Comparing Lenalidomide With Low Dose Dexamethasone Versus Lenalidomide in Second Line Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Hareth Nahi, MD, PhD, clinical assoc.professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI-RV-MM-10-07/ RV-MM-PI 0627; 2010-021857-38 (EudraCT Number)
Record Dates: First submitted 2011-09-07; First posted 2011-10-12 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Myeloma
Keywords: Relapsed and refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Revlimid (Experimental)
  Interventions: Drug: Revlimid
- Revlimid and dexamethasone (No Intervention)

INTERVENTIONS:
Drug: Revlimid — Group R:25 mg lenalidomide 21 of 28 days will be given orally as maintenance .
  Arms: Revlimid

SUMMARY:
This is:

* A prospective, randomized, open, phase II, multi-centre, interventional study. Patients who are in at least PR and have received lenalidomide as 2nd line treatment for MM will be recruited.
* The patients will be randomized into two groups. Group R will receive lenalidomide 25 mg/day p.o. continuously for 21 days and group Rb will receive a similar dose of lenalidomide with the addition of 40 mg of dexamethasone p.o. on days 1, 8, 15 and 22 of every 28 day treatment cycle. Study includes a maximum of 24 cycles including two consolidating cycles per patients.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria - all subjects must:

1. Be at least 18 years of age
2. Subjects must have a documented diagnosis of MM and have either refractory or relapsed and refractory after first line treatment disease defined as:

   * Primary refractory
   * Refractory
   * Relapsed and Refractory
3. Subjects must have undergone prior treatment with one treatment line of anti-myeloma therapy. Induction therapy followed by ASCT and consolidation/maintenance will be considered as one line.Have a confirmed diagnosis of MM
4. Have received lenalidomide after one prior treatment for MM and have reached at least a partial response (PR), according to IMWG criteria, including two consolidating cycles. Subjects have experienced a response at least PR after starting treatment with lenalidomide and cortisone cycles.
5. Have personally signed and dated a legally effective written informed consent form prior to admission to the study.
6. Must be willing and able to understand and comply with the study requirements.
7. Females of childbearing potential must agree to ongoing pregnancy testing and to practice contraception.
8. Male must agree to practice contraception

Exclusion Criteria:

1. Any of the following laboratory abnormalities:

   * Absolute neutrophil count (ANC) < 1,000/µL
   * Platelet count < 75,000/ µL
   * Creatinine Clearance < 45 mL/min according to Cockcroft-Gault formula
   * Serum SGOT/AST or SGPT/ALT > 3.0 x upper limit of normal (ULN)
   * Serum total bilirubin > 2.0 mg/dL
2. ECOG performance status <4.
3. Individuals who have had a stem-cell transplant as a 2nd line treatment for MM
4. Individuals who have taken any experimental drugs or participated in a clinical trial within 30 days prior to screening.
5. Individuals with significant psychiatric illness or a clinically significant acute/chronic uncontrolled medical condition that might affect their experience of myeloma symptoms or their ability to describe them.
6. Pregnant or lactating females.
7. Any other clinically significant medical disease or condition that, in the Investigator´s opinion, may interfere with protocol adherence or a subject´s ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-03; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Time to progression | 24 months

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | participants will be followed for the duration of hospital stay, an expected average of 2 years
  Number of Participants with Adverse Events

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Karolinska Inst., Stockholm
  - Karolinska Institute, Stockholm

REFERENCES:
- [Derived] Lund J, Gruber A, Lauri B, Duru AD, Blimark C, Swedin A, Hansson M, Forsberg K, Ahlberg L, Carlsson C, Waage A, Gimsing P, Vangsted AJ, Frolund U, Holmberg E, Gahrton G, Alici E, Hardling M, Mellqvist UH, Nahi H. Lenalidomide versus lenalidomide + dexamethasone prolonged treatment after second-line lenalidomide + dexamethasone induction in multiple myeloma. Cancer Med. 2018 Jun;7(6):2256-2268. doi: 10.1002/cam4.1422. Epub 2018 Apr 19. PMID 29673108